CLINICAL TRIAL: NCT02489292
Title: Prospective, Open Label, Multicenter, Efficacy and Safety Study of Several Infusions of HepaStem in Urea Cycle Disorders Paediatric Patients
Brief Title: Study to Evaluate the Efficacy of HepaStem in Urea Cycle Disorders Paediatric Patients (HEP002)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cellaion SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEP002
Record Dates: First submitted 2014-11-06; First posted 2015-07-03 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Urea Cycle Disorders
Keywords: Urea Cycle Disorder; UCD; cell therapy; stem cell
MeSH Terms: conditions — Urea Cycle Disorders, Inborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HepaStem (Experimental): Target total dose 50x10E6 cells/kg
  Interventions: Biological: HepaStem

INTERVENTIONS:
Biological: HepaStem — HepaStem will be administered in maximum 4 infusion days, spread over an 8-week period with an interval of 2 to 3 weeks between infusion days. The target total dose of cells will be 50x10E6 cells/kg body weight

SUMMARY:
The aim of the study is to assess the efficacy of HepaStem treatment in paediatric patients suffering from urea cycle disorders.

ELIGIBILITY:
Main Inclusion Criteria:

* Paediatric patients < 12 years prior to infusion
* Patient presents with UCD
* Patient shows patency of the portal vein and branches, with normal flow velocity as confirmed by Doppler US and accessibility of the portal vein and /or affluants.

Main Exclusion Criteria:

* Patient has mild disease severity, easily controlled under standard of care therapy, with no recurrent metabolic crises.
* Patient is registered on a liver transplant waiting list or is scheduled for living donor liver transplantation before the end of the study.
* Patient presents acute liver failure.
* Patient presents clinical or radiological evidence of liver cirrhosis.
* Patient presents or has a history of hepatic or extrahepatic malignancy.
* Patient has a known clinically significant cardiac malformation.
* Patient has a personal history of venous thrombosis, or has a clinically significant abnormal value for protein S, protein C, anti-thrombin III, and /or activated Protein C Resistance (aPCR) at screening. In case of known family history, a complete coagulation work-up should be performed. In all above described cases, results need to be discussed with PB before enrolling the patient in the study.
* Patient had or has a renal insufficiency treated by dialysis.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Efficacy as determined by de novo ureagenesis (C13 tracer method) | at 6m post-first infusion day

SECONDARY OUTCOMES:
Efficacy as determined by de novo ureagenesis (C13 tracer method) | at 3, 9 and 12 months post-first infusion day
Efficacy as determined by Ammonia (NH3) values | up to 12 months post-first infusion day
Efficacy as determined by amino acids in plasma | up to 12 months post-first infusion day
Efficacy as determined by report of metabolic decompensations | up to 12 months post-first infusion day
Efficacy as determined by report on actual supportive treatment, adjustment of protein restriction and amino acids supplements | up to 12 months post-first infusion day
Efficacy as determined report on behavior, cognitive skills and health-related quality-of-life indicators | up to 12 months post-first infusion day
To evaluate the safety during the year following HepaStem infusions (composite) | up to 12 months post-first infusion day
  Safety evaluation in terms of (1) clinical status, (2) portal vein hemodynamics, (3) morphology of the liver, bile ducts and portal system, (4) laboratory tests, (5) De novo detection of donor-specific circulating anti-human leukocyte antigen (HLA) antibodies, and/or other immune-related markers, (6) serious adverse events and clinically significant adverse events related to HepaStem, technical intervention, and concomitant treatments.

CONTACTS AND LOCATIONS:
Locations (6):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Hôpital Jeanne de Flandre, CHRU Lille, Lille, France
- Instytut - Pomnik Centrum Zdrowia Dziecka, Warsaw, Poland
- Spain (3):
  - Hospital Materno Infatil de Badajoz, Badajoz
  - Hospital Universitari Vall d'Hebron de Barcelona, Barcelona
  - Hospital Materno Infantil de Málaga, Málaga